CLINICAL TRIAL: NCT01265199
Title: Phase I Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Properties of Oral AT-406 in Combination With Daunorubicin and Cytarabine in Patients With Poor-risk, Acute Myelogenous Leukemia (AML)
Brief Title: Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Properties of Oral AT-406 in Combination With Daunorubicin and Cytarabine in Patients With Poor-risk Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated before a MTD was determined for administrative reasons
Sponsor: Ascenta Therapeutics (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-406-CS-002
Record Dates: First submitted 2010-12-20; First posted 2010-12-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myelogenous Leukemia (AML)
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide; Daunorubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AT-406 in combination with daunorubicin and cytarabine — Oral AT-406 (capsule) given once daily on days 1-5 of induction therapy with daunorubicin 90 mg/m2 I.v. on days 1-3 and cytarabine 100 mg/m2 i.v. by continuous infusion on days 107 of induction therapy.

SUMMARY:
The main purpose of this study are to determine the maximum dose of AT-406 that can be safely given in combination with cytarabine and daunorubicin to humans. Other purposes are to determine how the drug is broken down in the body, and to see if there are any molecular interactions that can help determine how AT-406 works. Side effects will also be studied in an effort to make sure that this drug is safe to take.

DETAILED DESCRIPTION:
This is an open label, multi-center, dose escalation study to determine the MTD of oral AT-406 combined with daunorubicin and cytarabine in patients with poor-risk AML. Treatment with AT-406 will be administered to up to 60 patients at approximately 7 investigational sites in the US. Patients will be enrolled in open label sequential cohorts of up to 12 patients to determine the MTD of AT-406 in combination with daunorubicin and cytarabine. Dose finding will occur during the induction cycle of the regimen. AT-406 will not be administered in consolidation cycles. Patients who require re-induction during initial treatment will be removed from the study and replaced (if needed) in order to assess at least 3 evaluable patients at each dose level.

Clinical and laboratory parameters will be assessed to evaluate the toxicity of AT-406. In addition, pharmacokinetic (PK) and pharmacodynamic (PDy) blood samples will be analyzed for plasma concentrations and PDy effect of AT-406, respectively.

ELIGIBILITY:
Eligibility Criteria:

Inclusion:

* Male or females patients ages 18 to 74
* Morphological diagnosis of untreated or relapsed non-M3 AML according to WHO diagnostic criteria who exhibit at least one poor-risk feature and are not be known to exhibit any favorable cytogenetic features or variants.
* Patients with relapsed AML and patients with prior autologous or allogeneic hematopoietic stem cell transplantations are eligible if relapse occurred following a remission of ≥ 6 months.
* Patients must have an ECOG score of ≤ 2,
* Adequate cardiac, liver and renal function.

Exclusion:

* Must not have any evidence of CNS leukemia.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine Number of Participants with Adverse Events as a Measure of Safety and Tolerability of oral AT-406 in combination with daunorubicin and cytarabine. | 15 months
  Determine Number of Participants with Adverse Events as a Measure of Safety and Tolerability of AT-101.

SECONDARY OUTCOMES:
Determine the pharmacokinetic profile of AT-406 and daunorubicin and cytarabine | 15 months
  To determine how the drug is absorbed, distributed, metabolized, and eliminated by the body.

CONTACTS AND LOCATIONS:
Overall Officials: J. Mel Sorensen, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (6):
- United States (6):
  - Univerity of Chicago, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University at St. Louis Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University at Jeanes Hospital, Philadelphia, Pennsylvania